CLINICAL TRIAL: NCT00208013
Title: The Survey About Resting Metabolic Rate and Its Related Factors in Terminal Patients
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Wen-Yuan, Lin, China Medical University Hospital
Other Study IDs: 94-2314-B-039-025
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2005-07

CONDITIONS: Advanced Cancers
Keywords: resting energy expenditure; cachexia; advanced cancer; advanced cancer patients
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cachectic patients often lose their appetite, lose weight, and are prone to weakness and even death in advanced illness. Nutrition therapy is important and of concern to the investigators in cancer patients. More than 80% of terminal cancer or advanced illness patients get cachexia. Cachexia is a complex, multifactorial syndrome that results from a reduction in food intake, a variety of metabolic abnormalities (including hypermetabolism) or more often a combination of the two. Cachexia will progress with disease progression. Cachexia or weight loss is often the major cause of death or poor quality of life.

The change of resting energy expenditure (REE) is different in various tumor types. Most experts agree that the REE will increase in cancer cachexia syndrome. The more weight loss, the more cachexia will occur.

Overnutrition is not beneficial in terminal patients according to the Chiu and Easson studies. As the investigators know, few studies focus on REE in terminal patients. In this study, samples are from a hospice palliative ward or from hospice home care patients in a medical center in mid-Taiwan. About 100 patients will be recruited. The investigators will analyze the relationship between REE and its related factors. After finishing the study, they will provide more evidence for treating cachexia in terminal patients.

DETAILED DESCRIPTION:
According to data from the Taiwanese government, cancer mortality has been the leading cause of death in Taiwan since 1982. The trend is increasing day by day. As the people are aging in Taiwan, the incidence of cancer will increase and it will be more important than before.

Cachectic patients often lose their appetite, lose weight, and are prone to weakness and even death in advanced illness. Nutrition therapy is important and of concern to the investigators in cancer patients. More than 80% of terminal cancer or advanced illness patients get cachexia. Cachexia is a complex, multifactorial syndrome that results from a reduction in food intake, a variety of metabolic abnormalities (including hypermetabolism) or more often a combination of the two. Cachexia will progress with disease progression. Cachexia or weight loss is often the major cause of death or poor quality of life.

The change of resting energy expenditure (REE) is different in various tumor types. Most experts agree that the REE will increase in cancer cachexia syndrome. The more weight loss, the more cachexia will occur.

Overnutrition is not beneficial in terminal patients according to the Chiu and Easson studies. As the investigators know, few studies focus on REE in terminal patients. In this study, samples are from a hospice palliative ward or from hospice home care patients in a medical center in mid-Taiwan. About 100 patients will be recruited. The investigators will analyze the relationship between REE and its related factors. After finishing the study, they will provide more evidence for treating cachexia in terminal patients.

ELIGIBILITY:
Inclusion Criteria:

* Terminal cancer patients who were admitted to a hospice palliative ward in one medical center located in mid-Taiwan

Exclusion Criteria:

* Patient could not complete the examination of resting metabolic rate using MedGerm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: advanced cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yuan Lin, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- CMUH, Taichung, Taiwan